CLINICAL TRIAL: NCT06363409
Title: The Acute and Accumulative Effects of Almonds on Exercise Recovery
Brief Title: The Acute and Accumulative Effects of Snack Foods on Exercise Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-1353
Record Dates: First submitted 2024-04-02; First posted 2024-04-12 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Muscle Strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cereal bar arm (Experimental): weight lifting exercise and post-exercise cereal bar consumption
  Interventions: Other: Cereal Bar as a recovery food snack
- Almond arm (Experimental): weight lifting exercise and post-exercise almond consumption
  Interventions: Other: Almond

INTERVENTIONS:
Other: Cereal Bar as a recovery food snack — Cereal bar as a recovery snack food
  Arms: Cereal bar arm
Other: Almond — Almond as a recovery snack food
  Arms: Almond arm

SUMMARY:
The purpose of the research is two-fold. One goal is to determine if post-exercise almond or cereal bar consumption can promote muscle gain as well as increasing muscular strength throughout an eight-week weight training program. The other goal is to assess the short-term effects of almonds or cereal bar on recovery that may explain the overall long-term adaptations.

ELIGIBILITY:
Inclusion Criteria:

* BMIs of 18.5-30 kg/m2
* participate in no more than 3 hours of structured exercise per week

Exclusion Criteria:

* weight training more than 30 min/week,
* smoking,
* use of medications known to impact inflammation,
* musculoskeletal limitations,
* use of supplements within 1 month of participation that are known to impact body composition, antioxidant or inflammatory status,
* regular consumption of more than 2 servings of nuts per week,
* unwillingness to refrain from recovery treatments during the study such as hydrotherapy, massage, stretching, compression garments, anti-inflammatory medications and topical applications.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
delayed onset of muscle soreness | baseline, 24 hour, 48 hour, and 72 hour after baseline
  measuring delayed onset of muscle soreness using visual analogue scale (VAS)
markers of muscle damage | Baseline, 24 hour, 48 hour and 72 hour after baseline
  Blood markers of muscle damage (creatine kinase (u/L))
changes in strength | Baseline and 8 weeks
  muscle cross-sectional area of the calf via peripheral quantitative computerized tomography (pQCT)
changes in body composition | Baseline and 8 weeks
  measuring body composition by dual energy x-ray absorptiometry (DXA)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kern, PhD, RD, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No